CLINICAL TRIAL: NCT01083108
Title: Effects of Caloric Restriction Alone Versus Postoperative Caloric Restriction Following Bariatric Surgery on Glucose Metabolism in Patients With Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 100064; 10-DK-0064
Record Dates: First submitted 2010-03-06; First posted 2010-03-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12-13

CONDITIONS: Obesity; Bariatric Surgery; Morbid Obesity; Diabetes Mellitus Type 2; Diet Therapy
Keywords: Behavioral Weight Loss Treatment; Bariatric Surgery; Diabetes Type II; Obesity; Adult; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass; Caloric Restriction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical Arm (Active Comparator): Low-calorie Diet
  Interventions: Other: Caloric Restriction
- Surgical Arm (Experimental): Roux-en-Y Gastric Bypass
  Interventions: Other: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Other: Roux-en-Y Gastric Bypass — The surgical group will be studied before and 6 days after bariatric surgery.
  Arms: Surgical Arm
Other: Caloric Restriction — The non-surgical group will be studied before and after receiving a hypocaloric diet for 6 days mimicking the typical postoperative diet.
  Arms: Non-surgical Arm

SUMMARY:
Background:

* Bariatric surgery is the most effective way to achieve significant, long-term weight loss. It has also been shown to be an effective therapy for obese individuals with type 2 diabetes: more than 70 percent of patients no longer need medications for diabetes after surgery. This resolution of diabetes is predominately caused by marked weight loss resulting in improved insulin sensitivity. However, the beneficial effects of bariatric surgery on type 2 diabetes cannot be accounted for entirely by weight loss, because many bariatric surgery patients have resolution of diabetes within 1 week following bariatric surgery, even before they lose a clinically significant amount of weight.
* One possible reason for the rapid resolution of diabetes after bariatric surgery .is that during the first week after surgery, patients can eat very little (about 300 Calories per day). It is well known that reducing calories to this level improves diabetes. Another possibility is that changes in the flow of food through the intestines may improve diabetes. Evidence for this comes from the observation that patients after gastric bypass have better glucose levels than those who have gastric banding. Researchers are interested in determining how much of the improvement in diabetes in the first week after Roux-en-Y gastric bypass (RYGBP) surgery is due to restricting calories, and how much is due to other factors, such as bypassing the upper part of the small intestine.

Objectives:

* To determine the change in total body insulin sensitivity after RYGBP compared to caloric restriction without surgery.
* To study possible reasons for improvements in diabetes after RYGBP.

Eligibility:

- Individuals 18 to 60 years of age who have a body mass index (BMI) greater than 35 and have type 2 diabetes.

Design:

- This is not a randomized study, and patients will not receive bariatric surgery as part of this study.

Two groups of patients will be studied: those scheduled for RYGBP surgery and those not undergoing surgery.

* RYGBP Surgery Participants:
* Up to 3 weeks before surgery, participants will spend 2 nights and days at the Vanderbilt University Clinical Research Center or the NIH Clinical Center for testing to learn about how their bodies handle sugar and use energy. During the 5 days prior to these tests, participants will be asked to not take diabetes medications, and will check blood sugar at least twice a day.
* From 8 days before surgery, participants will begin an 800 Calorie per day liquid diet to prepare for surgery.
* After surgery and discharge, participants will be readmitted to the Clinical Research Center at Vanderbilt or NIH for further tests and diet monitoring. Diabetes medications may be adjusted or stopped altogether based on the results of the tests.
* Non-surgery Participants:
* Participants will spend 2 nights and days in the NIH Clinical Center for testing to learn about how their bodies handle sugar and use energy. During the 5 days prior to these tests, participants will be asked to not take diabetes medications, and will check blood sugar at least twice a day.
* After the tests, participants will begin an 800 Calorie per day liquid diet for 8 days.
* After 8 days, participants will be readmitted to the Clinical Center at NIH for 1 week of further tests and a 300 Calorie per day diet. Diabetes medications may be adjusted or stopped altogether based on the results of the tests.

DETAILED DESCRIPTION:
Background

Presently it is unknown whether the rapid normalization of glucose metabolism in obese patients with type 2 diabetes after bariatric surgery (before major weight loss occurs) is primarily due to acute postoperative caloric restriction or due to changes in intestinal effects on insulin secretion and sensitivity. We speculate that bypassing the stomach and proximal small intestine affects glucose metabolism beyond simple caloric restriction, and that the mechanisms are related to changes in hepatic and muscle insulin sensitivity, changes in vagal afferent signals, and changes in incretins and other gut hormones.

Aim

To compare the effects of pure caloric restriction with caloric restriction early after bariatric surgery (Roux-en-Y Gastric Bypass, RYGBP) in patients with type 2 diabetes, and to investigate the mechanisms that explain the observed difference in glucose metabolism

Methods

In patients with type 2 diabetes we will study the short-term changes in glucose metabolism, insulin sensitivity and gut hormone levels using a parallel group design. The non-surgical group will be studied before and after receiving a hypocaloric diet for 6 days mimicking the typical postoperative diet. The surgical group will be studied before and 6 days after bariatric surgery. The primary outcome will be the change in total body insulin sensitivity attributable to caloric restriction alone versus caloric restriction after RYGBP. Non-surgical subjects studied at NIH may enter an optional long-term weight loss phase.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Clinical diagnosis of Type 2 diabetes mellitus
  2. Age 18-60 years
  3. Body mass index greater than or equal to 35 kg/m(2)
  4. Either

     --a. Patients scheduled for Roux-en-Y gastric bypass at Vanderbilt University Medical Center or University of Maryland

     OR

     --b. Patients matched for race, sex, BMI (plus or minus 15%), and age (plus or minus 5 years) to RYGBP patients, above, but NOT scheduled for bariatric surgery.
  5. Subjects must have an endocrinologist or primary care provider who manages their diabetes.

EXCLUSION CRITERIA:

1. Current use of insulin
2. Use of exenatide, sitagliptin (or other dipeptidyl peptidase inhibitor), thiazolidinediones, or experimental diabetes medication within the past 3 months
3. Medical condition that alters glucose metabolism (other than type 2 diabetes) or weight (e.g. chronic inflammatory diseases, monogenic obesity, Prader-Willi syndrome)
4. Current use of medication that alters glucose metabolism (other than oral diabetes medications) or weight (e.g. corticosteroids, atypical antipsychotic drugs)
5. Significant comorbidity that, in the opinion of the investigators, will increase risk to the subject, (e.g. current treatment for cancer, renal failure)
6. Positive urine pregnancy test or plans to become pregnant during the clinical trial
7. Psychiatric or cognitive disorder that will, in the opinion of the investigators, limit the subject's ability to comply with study procedures
8. Body weight greater than 450 lbs
9. History of previous bariatric surgical procedure or other surgery altering the length or arrangement of the intestines (e.g. Whipple procedure)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03-31; Primary Completion 2013-05-22 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is the change in total body insulin sensitivity due to RYGBP alone using the euglycemic hyperinsulinemic clamp technique. | 2 years
  Insulin sensitivity will be determined using the gold standard euglycemic hyperinsulinemic clamp method, which directly measures total body insulin sensitivity as the glucose disposal rate, M, during steady state conditions of euglycemia and hyperinsulinemia. A two- stage clamp will be performed, using first a low-dose insulin infusion (to determine hepatic insulin sensitivity), followed by a high-dose insulin infusion (to determine muscle insulin sensitivity).

SECONDARY OUTCOMES:
The secondary outcomes are changes in insulin sensitivity, insulin secretion, and gut hormones due to caloric restriction alone, caloric restriction plus RYGBP, and RYGBP alone. | 2 years
  In addition to assessing total body insulin sensitivity, we will evaluate hepatic insulin sensitivity, insulin secretion and gut hormones for threeconditions:1. Diet alone (Before vs. after 6 day caloric restriction in the non-surgical group)2. Diet plus bariatric surgery (Before vs. after 6 day caloric restriction and surgery in the RYGBP group)3. Bariatric surgery alone (After 6 day caloric restriction in RYGBP group vs. non-surgical group)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina I Rother, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (3):
- United States (3):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Butler AE, Janson J, Bonner-Weir S, Ritzel R, Rizza RA, Butler PC. Beta-cell deficit and increased beta-cell apoptosis in humans with type 2 diabetes. Diabetes. 2003 Jan;52(1):102-10. doi: 10.2337/diabetes.52.1.102. PMID 12502499
- [Background] Meier JJ, Bhushan A, Butler AE, Rizza RA, Butler PC. Sustained beta cell apoptosis in patients with long-standing type 1 diabetes: indirect evidence for islet regeneration? Diabetologia. 2005 Nov;48(11):2221-8. doi: 10.1007/s00125-005-1949-2. Epub 2005 Oct 5. PMID 16205882
- [Background] Turner RC, Cull CA, Frighi V, Holman RR. Glycemic control with diet, sulfonylurea, metformin, or insulin in patients with type 2 diabetes mellitus: progressive requirement for multiple therapies (UKPDS 49). UK Prospective Diabetes Study (UKPDS) Group. JAMA. 1999 Jun 2;281(21):2005-12. doi: 10.1001/jama.281.21.2005. PMID 10359389